CLINICAL TRIAL: NCT01797250
Title: Neonatal and Pediatric Studies Using a Bedside Respiratory Patient Monitoring System With the Functional Patient Monitoring PCBA-1
Brief Title: Pulse Oximetry_Performance Testing- PCBA-1 (Printed Circuit Board Assembly) NEO/PEDS
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0308
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Subjects With an Existing Intra-arterial Line

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine accuracy specifications of the pulse oximeter in the NEO/PEDS subject population

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal guardian is willing and able to sign informed consent prior to study initiation.
2. Subject is able to participate for the duration of the evaluation. In most instances, the length of the study will not exceed twenty-four hours.
3. Subject satisfies a specified sensor requirement (see Table 1).
4. Requires use of an intra-arterial line for medical reasons such as continuous blood pressure monitoring or frequent arterial blood draws.
5. Subject is able to accommodate multiple sensors.
6. Neonatal subjects up to 1 month of age or Pediatric subjects 1 month up to 18 years old.

Exclusion Criteria:

1. Subjects that have an existing health condition, in which the investigators determine that safe or accurate oximetry measures may not be obtained at the areas where the pulse oximetry sensor could be placed, will not be included in the study. For example, anyone with burns, abrasions or surface lesions on the contact areas would be excluded.
2. Any subject whose treatment or condition would be compromised if they were to participate in this study and any patient whose use of a pulse oximeter and sensor would present a potential for serious risk to health, safety, or welfare.
3. Subject has severe contact allergies that may react to standard adhesive materials found in pulse oximetry sensors.
4. Subject cannot be reliably monitored with a pulse oximeter as a result of inadequate pulsatile signals.
5. Subject has had a procedure using injected intravascular dyes within 24 hours preceding testing

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will include male and female pediatric and neonatal patients who meet the specified sensor weight requirements with an existing intra-arterial line, typically found in hospital intensive care areas. Subjects of all racial and ethnic backgrounds may be included in the studies.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
SpO2 Accuracy (percentage of blood oxygen saturation) | Planned duration of study was up to 12 months. Duration of subject participation: 1-24 hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital- Los Angeles, Los Angeles, California
  - Wasatch Neonatal, Orem, Utah